CLINICAL TRIAL: NCT03180840
Title: Phase 3 Open-Label Switch Over Study to Assess Safety, Efficacy & PK of Pegunigalsidase Alfa (PRX-102) 2mg/kg IV Every 4 Weeks for 52 Weeks in Fabry Disease Patients Currently Treated With Enzyme Replacement Therapy Fabrazyme® or Replagal™
Brief Title: Safety, Efficacy, & PK of PRX-102 in Patients With Fabry Disease Administered Intravenously Every 4 Weeks
Acronym: BRIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protalix (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-102-F50
Record Dates: First submitted 2017-05-29; First posted 2017-06-08 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Fabry Disease
Keywords: Enzyme-Replacement Therapy; pegunigalsidase alfa; Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Intervention Model Description: Switch over study in patients previously receiving either agalsidase alfa or agalsidase beta and switched to pegunigalsidase alfa (PRX-102) for the treatment of Fabry disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegunigalsidase alfa (Experimental): Pegunigalsidase alfa 2 mg/kg intravenous infusion every 4 weeks
  Interventions: Biological: Pegunigalsidase alfa

INTERVENTIONS:
Biological: Pegunigalsidase alfa — Pegunigalsidase alfa 2 mg/kg every 4 weeks
  Other Names: PRX-102; Recombinant human alpha galactosidase-A

SUMMARY:
This open-label switchover study will assess the safety, efficacy, and pharmacokinetics of pegunigalsidase alfa (PRX-102) 2 mg/kg administered every 4 weeks for 52 weeks in Fabry patients previously treated with ERT: agalsidase alfa or agalsidase beta for at least 3 years. Safety and efficacy exploratory endpoints will be evaluated throughout the study period and pharmacokinetics will be obtained on Day 1 and Week 52.

DETAILED DESCRIPTION:
This is an open-label switchover study to assess the safety, efficacy, and pharmacokinetics of pegunigalsidase alfa treatment of 2 mg/kg every 4 weeks in patients previously treated with enzyme-replacement therapy (ERT): agalsidase alfa or agalsidase beta, for at least 3 years and on a stable dose (>80% labelled dose/kg) for at least the last 6 months. Following screening, patients will be enrolled and switched from their current ERT to receive intravenous (IV) infusions of pegunigalsidase alfa 2 mg/kg every 4 weeks for 52 weeks (total of 14 infusions). At the time of enrollment, premedication, if used for the agalsidase alfa or agalsidase beta infusions before enrollment, will be continued using the same premedication regimen during the first infusion with pegunigalsidase alfa and then will be gradually tapered down at the Investigator's discretion during the next infusions based on protocol-specified criteria. First infusions of pegunigalsidase alfa will be administered under controlled conditions at the investigation site. Based on the protocol-specified criteria, patients will be able to receive their pegunigalsidase alfa infusions at a home care setup once the Investigator and Sponsor Medical Monitor agree that it is safe to do so. Safety and efficacy exploratory endpoints will be assessed throughout the 52-week study. In the case of clear clinical deterioration, the treatment may be changed to 1.0 mg/kg every 2 weeks at the Investigator's discretion and discussion with the Medical Monitor.

ELIGIBILITY:
Key inclusion criteria:

Eligible subjects must fulfill the following inclusion criteria:

1. Age: 18-60 years
2. A documented diagnosis of Fabry disease
3. Males: plasma and/or leucocyte alpha galactosidase activity (by activity assay) less than lower limit of normal according to the laboratory reference ranges and one or more of the characteristic features of Fabry disease

   1. Neuropathic pain
   2. Cornea verticillata
   3. Clustered angiokeratoma
4. Females: historical genetic test results consistent with Fabry mutations, or in the case of novel mutations a first-degree male relative with Fabry disease, and one or more of the characteristic features of Fabry disease

   1. Neuropathic pain
   2. Cornea verticillata
   3. Clustered angiokeratoma
5. Treatment with agalsidase alfa or agalsidase beta for at least 3 years and on a stable dose (>80% labelled dose/kg) for at least last 6 months
6. eGFR ≥ 30 mL/min/1.73m^2 by CKD-EPI equation at screening visit
7. Availability of at least 3 historical serum creatinine evaluations since starting agalsidase alfa or agalsidase beta treatment and not more than 2 years old
8. Female patients and male patients whose co-partners are of child-bearing potential agree to use a medically accepted, highly effective method of contraception. These include combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, or sexual abstinence
9. Patients whose clinical condition, in the opinion of the Investigator, is suitable for treatment with ERT every 4 weeks.

Key exclusion criteria:

The presence of any of the following excludes a subject from study enrollment:

1. History of anaphylaxis or Type 1 hypersensitivity reaction to agalsidase alfa or agalsidase beta
2. History of renal dialysis or transplantation
3. Linear negative slope of eGFR of ≥ 2 mL/min/1.73m^2/year based on at least 4 serum creatinine values over approximately 2 years (including the value obtained at the screening visit)
4. History of acute kidney injury in the 12 months prior to screening, including specific kidney diseases (e.g., acute interstitial nephritis, acute glomerular and vasculitic renal diseases); non-specific conditions (e.g., ischemia, toxic injury); as well as extrarenal pathology (e.g., prerenal azotemia and acute post renal obstructive nephropathy)
5. Angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) therapy initiated or dose changed in the 4 weeks prior to screening
6. Urine protein to creatinine ratio (UPCR) at screening > 0.5 g/g or mg/mg or 500 mg/g and not treated with an ACE inhibitor or ARB
7. Females who are pregnant, planning to become pregnant during the study, or are breast feeding
8. Cardiovascular event (myocardial infarction, unstable angina) in the 6-month period before screening
9. Cerebrovascular event (stroke, transient ischemic attack) in the 6-month period before screening
10. Presence of any medical, emotional, behavioral, or psychological condition that, in the judgment of the Investigator and/or Medical Director, would interfere with the patient's compliance with the requirements of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - UAB Medicine, Birmingham, Alabama
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Infusion Associates, Grand Rapids, Michigan
  - Institute of Metabolic Disease, Dallas, Texas
  - University of Utah Hospital & Clinics, Salt Lake City, Utah
  - O & O Alpan, Fairfax, Virginia
- UZ Antwerpen, Edegem, Belgium
- Fakultní poliklinika Všeobecné fakultní nemocnice v Praze, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- Azienda Ospedaliera Universitaria "Federico II", Napoli, Italy
- Helse Bergen HF Haukeland Universitetssykehus, Bergen, Norway
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - The Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azimpour K, Dorling P, Koulinska I, Kunduri S, Lan Z, Poritz J, Tremblay G, Raad-Faherty A. Health State Utility Values in Fabry Disease: Insights from the Pegunigalsidase Alfa Clinical Trials. Adv Ther. 2025 Mar;42(3):1421-1434. doi: 10.1007/s12325-024-03095-2. Epub 2025 Jan 23. PMID 39847314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were treated with agalsidase beta or agalsidase alfa for at least three years and have been on a stable dose (>80% labelled dose/kg) for at least 6 months.
Pre-assignment Details: Screening details:
  A total of 52 patients were screened of whom 30 patients (24 males and 6 females) were enrolled and switched from agalsidase alfa or agalsidase beta to pegunigalsidase alfa over a 52-week period, of whom 29 patients (23 males and 6 females) completed the study.
Groups:
- Pegunigalsidase Alfa: Pegunigalsidase alfa 2.0 mg/kg intravenous infusion every 4 weeks for 12 months
Period: Overall Study
Arm/Group | Pegunigalsidase Alfa
Started | 30
Completed (Of the 30 patients who were enrolled in the study and treated,1 patient withdrew consent after receiving the first infusion of PRX-102 2.0 mg/kg and 29 patients completed the study. The PRX-102 dosing regimen was changed to 1.0 mg/kg E2W for 1 patient during the study. A further patient was treated for more than 52 weeks due to the COVID-19 pandemic restrictions.) | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose (partial or complete) of pegunigalsidase alfa in the study.
Arm/Group | Pegunigalsidase Alfa
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 2
  United States | 18
  Norway | 1
  Denmark | 1
  United Kingdom | 2
  Italy | 3
  Czechia | 3
Previous Enzyme Replacement Therapy (ERT) [Count of Participants; unit: Participants] — Previously treated with agalsidase beta or agalsidase alfa
  Participants
    Agalsidase alfa | 7
    Agalsidase beta | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events (TEAE) as Assessed by CTCAE v4.03
Description: Results represent the number of treatment-emergent adverse events (TEAE) that were considered possibly, probably, or definitely related to treatment.
Time Frame: Month 12
Measure: Number; unit: participants
Groups:
- PRX-102: Pegunigalsidase alfa 2.0 mg/kg intravenous infusion every 4 weeks for 12 months
Arm/Group | PRX-102
Number analyzed (Participants) | 30
participants
  At least 1 TEAE | 27
  At least 1 mild or moderate TEAE | 26
  At least 1 severe TEAE | 2
  At least 1 serious TEAE | 2
  At least 1 non-serious TEAE | 26
  At least 1 related TEAE | 9
  At least 1 related mild or moderate | 9
  At least 1 related severe TEAE | 0
  At least 1 related serious TEAE | 0
  At least 1 TEAE leading to withdrawal | 0
  At least 1 TEAE leading to death | 0

2. Other Pre Specified Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR was calculated based on the serum creatinine values that were assessed at Day 1, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 according to the CKD-EPI formula, baseline and Month 12 (week 52) reported. The change in eGFR from baseline measurement at Day 1 prior to first PRX-102 infusion to last measurement at Month 12 was summarized using descriptive statistics. The change was calculated for each subject and the reported value is the mean (Standard Error) of these changes.
Time Frame: Baseline and Month 12 (week 52)
Population: Any subjects who have at least one post-baseline observation.
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Groups:
- Efficacy Population: Number of Subjects Analysed
- Males: Number of Male Subjects Analysed
- Females: Number of Females Analysed
Arm/Group | Efficacy Population | Males | Females
Number analyzed (Participants) | 29 | 23 | 6
mL/min/1.73m^2
  Baseline | 99.44 (4.15) | 100.68 (4.96) | 94.69 (6.76)
  Month 12 (week 52) | 100.65 (3.14) | 103.24 (3.46) | 91.15 (6.39)
  Change from Baseline to Month 12 (week 52) | -1.27 (1.39) | -0.64 (1.57) | -3.54 (3.12)

3. Other Pre Specified Outcome: Plasma Lyso-Gb3
Description: Globotriaosylsphingosine (Lyso-Gb3) is Fabry disease specific biomarker that can assess treatment outcome, for which was measured at Baseline, weeks 12, 24, 40 and 52. The mean Plasma Lyso-Gb3 concentrations at baseline and Month 12 (week 52) and the mean change from Baseline reported.
  The change from baseline to month 12 was calculated for each subject and the reported values is the mean (Standard Error) of these changes.
Time Frame: Baseline and month 12 (Week 52)
Population: Any subjects who have at least one post-baseline observation.
Measure: Mean (Standard Error); unit: nM
Arm/Group | Efficacy Population | Males | Females
Number analyzed (Participants) | 29 | 23 | 6
nM
  Baseline | 19.36 (3.35) | 23.27 (3.82) | 4.35 (1.00)
  Month 12 (week 52) | 22.23 (3.60) | 27.05 (4.00) | 4.52 (1.10)
  Change from Baseline to Month 12 (week 52) | 3.01 (0.94) | 3.79 (1.14) | 0.17 (0.34)

4. Other Pre Specified Outcome: Quality of Life by EQ-VAS
Description: The EQ-VAS, of the EQ-5D-5L questionnaire, records the subject's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' (Score 100) and 'Worst imaginable health state' (Score 0). The change from baseline to month 12 was calculated for each subject and the reported value is the mean (Standard Error) of these changes.
Time Frame: Baseline and 12 months (week 52)
Population: Any subjects who have at least one post-baseline observation.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Efficacy Population
Number analyzed (Participants) | 29
scores on a scale
  Baseline | 78.3 (3.1)
  Month 12 (week 52) | 82.1 (2.9)
  Change from Baseline to Month 12 (week 52) | 3.0 (2.2)

5. Other Pre Specified Outcome: Pharmacokinetics - Cmax
Description: Pharmacokinetic (PK) parameters were derived from the plasma concentration versus time profiles. Cmax is the maximal plasma concentration of a drug after administration. Results reported represent the values following a single dosing of the study drug.
Time Frame: Day 1, Month 9 or 11, and Month 12
Population: All subjects who received at least one dose of PRX-102 and for whom a sufficient number of evaluable samples were available to determine at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Safety Population: Number of subjects analysed
Arm/Group | Safety Population
Number analyzed (Participants) | 30
ng/mL | 35876.7 (11942.2)

6. Other Pre Specified Outcome: Pharmacokinetics - AUC
Description: PK parameters were derived from the plasma concentration versus time profiles. AUC is the area under the plasma concentration curve from 0 hour to infinity. Results reported represent the values following a single dosing of the study drug.
Time Frame: Day 1, Month 9 or 11, and Month 12.
Population: All subjects who received at least one dose or PRX-102 and for whom a sufficient number of evaluable samples were available to determine at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Safety Population
Number analyzed (Participants) | 30
ng*hr/mL | 1797464.1 (822632.4)

7. Other Pre Specified Outcome: Pharmacokinetics - Terminal Half Life
Description: PK parameters were derived from the plasma concentration versus time profiles. t1/2 = half life. Results reported represent the values following a single dosing of the study drug.
Time Frame: Day 1, Month 9 or 11, and Month 12.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Safety Population
Number analyzed (Participants) | 30
hour | 100.1 (58.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment until 30 days following the final study dose, an average of 13 months.
Groups:
- All Patients: Analysis of AEs was performed on TEAEs, defined as AEs occurring after the start of the first infusion with pegunigalsidase alfa.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=30)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=30)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (17)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Headache (Nervous system disorders) | 3 (4)
Paraesthesia (Nervous system disorders) | 3 (3)
Neuralgia (Nervous system disorders) | 2 (2)
Pain (General disorders) | 3 (9)
Fatigue (General disorders) | 5 (6)
Chest discomfort (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7)
Gastroenteritis (Infections and infestations) | 2 (4)
Sinusitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Viral infections (Infections and infestations) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)

LIMITATIONS AND CAVEATS:
Small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial agreement provided to the sites and Investigators contains a Publication paragraph that indicates the following: shall not, without the Sponsor's prior written consent, independently publish, present or otherwise disclose any results of or information pertaining to the trial until a multi-center publication is published, subject to certain limitations regarding timing and the confidentiality of unpublished data.

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03180840/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03180840/SAP_001.pdf